CLINICAL TRIAL: NCT04430491
Title: Multi-center Validation of a Radiomics Based Model for the Diagnosis of Idiopathic Pulmonary Fibrosis
Brief Title: To Evaluate the Use of Radiomics to Classify Between Idiopathic Pulmonary Fibrosis and Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Other Study IDs: RESPIRE_2019
Record Dates: First submitted 2020-05-01; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Usual Interstitial Pneumonia
Keywords: Lung; CT; UIP; IPF; ILDs
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training dataset: No interventions
  Interventions: Diagnostic Test: radiomics
- Validation dataset: No interventions
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics — The high-throughput extraction of large amounts of quantitative image features from medical images

SUMMARY:
To investigate the ability of machine learning models based on radiomic features extracted from thin-section CT images to differentiate IPF patients from non-IPF interstitial lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* UIP with final diagnosis in biopsy
* ILDs with final diagnosis in biopsy

Exclusion Criteria:

* patients with no biopsy confirmation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the hospital for lung disease. Two cohorts were included. One from Belgium, and a second one from the US.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
IPF classifier | Up to 30 weeks
  Model based on Radiomic that can differentiate IPF from ILDs.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided